CLINICAL TRIAL: NCT07272031
Title: Randomized Controlled Trial to Evaluate the Effectiveness of Three Different 15-Minute Office Massage Types (Head, Cervical Area, Hand) on Autonomic Nervous System Balance and Chronic Stress Reduction Using Heart Rate Variability (HRV)
Brief Title: Office Massage Effects on HRV and Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riga Stradins University (Other)
Responsible Party: Principal Investigator, Una Veseta, Lead Researcher, Riga Stradins University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OM_HRV_2025_RCMC
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Occupational Health; Autonomic Nervous System (ANS) Functioning and Mood State; Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Head Massage (Active Comparator): Duration and Frequency: 15 minutes per session, 2 times per week for 4 consecutive weeks (8 sessions total). Focus: Massage focuses on the scalp, temples, and auricles (outer ear) with the aim of stimulating cranial nerves, particularly branches of the vagus nerve. The procedure is performed by a licensed massage therapist while the participant is seated in an office chair.
  Interventions: Procedure: Head Massage Intervention
- Cervical Area Massage (Active Comparator): Duration and Frequency: 15 minutes per session, 2 times per week for 4 consecutive weeks (8 sessions total). Focus: Deep tissue and kneading massage techniques applied primarily to the trapezius muscles, levator scapulae, and sub-occipital region (neck/shoulders). The procedure is performed by a licensed massage therapist while the participant is seated in an office chair.
  Interventions: Procedure: Cervical Area Massage Intervention
- Hand Massage (Active Comparator): Duration and Frequency: 15 minutes per session, 2 times per week for 4 consecutive weeks (8 sessions total). Focus: Compression, rubbing, and stroking techniques applied to the palmar and dorsal surfaces of the hands, fingers, and wrists. The procedure is performed by a licensed massage therapist while the participant is seated in an office chair.
  Interventions: Procedure: Hand Massage Intervention
- Quiet Rest Control (Placebo Comparator): Duration and Frequency: Participants are seated in the same office chair for a structured 15-minute period, 2 times per week for 4 consecutive weeks (8 sessions total). Focus: Participants are instructed to sit quietly, avoid work-related activity, and refrain from using electronic devices. This arm controls for the effect of researcher attention and time spent away from work.
  Interventions: Other: Quiet Rest Control

INTERVENTIONS:
Procedure: Head Massage Intervention — 15 minutes per session, 2 times per week for 4 consecutive weeks (8 sessions total). Focus: Massage focuses on the scalp, temples, and auricles (outer ear) with the aim of stimulating cranial nerves, particularly branches of the vagus nerve. The procedure is performed by a licensed massage therapist while the participant is seated in an office chair.
  Arms: Head Massage
Procedure: Cervical Area Massage Intervention — 15 minutes per session, 2 times per week for 4 consecutive weeks (8 sessions total). Focus: Deep tissue and kneading massage techniques applied primarily to the trapezius muscles, levator scapulae, and sub-occipital region (neck/shoulders). The procedure is performed by a licensed massage therapist while the participant is seated in an office chair.
  Arms: Cervical Area Massage
Procedure: Hand Massage Intervention — 15 minutes per session, 2 times per week for 4 consecutive weeks (8 sessions total). Focus: Compression, rubbing, and stroking techniques applied to the palmar and dorsal surfaces of the hands, fingers, and wrists. The procedure is performed by a licensed massage therapist while the participant is seated in an office chair.
  Arms: Hand Massage
Other: Quiet Rest Control — Participants are seated in the same office chair for a structured 15-minute period, 2 times per week for 4 consecutive weeks (8 sessions total). Focus: Participants are instructed to sit quietly, avoid work-related activity, and refrain from using electronic devices. This arm controls for the effect of researcher attention and time spent away from work.
  Arms: Quiet Rest Control

SUMMARY:
This study is a randomized controlled trial designed to investigate which of three short office massage types (head, neck/shoulder area, or hand) is most effective for reducing chronic stress in women who perform sedentary office work.

Many sedentary female office employees experience long-term tension and work-related strain, which can affect the body's ability to recover. The investigators are testing whether a 15-minute massage, performed twice a week for four weeks, can help restore balance within the body.

The investigators will evaluate the impact of these massages using Heart Rate Variability (HRV)-an objective measure that shows how well the body manages stress (autonomic nervous system balance)-as well as analyzing participants' self-reported levels of perceived stress, sleep quality, and overall well-being. Participants receiving massage will be compared to a control group engaging in quiet rest.

ELIGIBILITY:
Inclusion Criteria:

Biological females aged 18 years or older. Currently working in an office job with at least 75% of the working day spent sitting (sedentary work).

Must report a regular menstrual cycle (cycle length 21-35 days) for at least the past 6 months.

Able to attend all scheduled intervention sessions (8 sessions over 4 weeks). Able to provide informed consent to participate in the study.

Exclusion Criteria:

Use of hormonal contraceptives or other hormone-containing therapies (e.g., Intrauterine Device (IUDs), patches, birth control pills).

Pregnancy, current breastfeeding, or planning pregnancy during the study period.

Menopause (natural or surgically induced). Diagnosis of a severe chronic disease (e.g., heart failure, insulin-dependent diabetes, diagnosed neurological disorder).

Active cancer or history of cancer within the last 5 years. Current diagnosis of a major psychiatric disorder (e.g., major depressive disorder, bipolar disorder).

Current use of psychotropic medications that could significantly affect Heart Rate Variability (HRV) (e.g., certain beta-blockers, anti-depressants).

History of recent surgery (within the last 3 months) in the neck or upper extremities.

Participation in another clinical trial simultaneously.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Morning Resting Heart Rate Variability (rMSSD) at 4 Weeks | Baseline, Periprocedural and Week 4
Change from Baseline in Perceived Stress Level (PSS-10 Score) at 4 Weeks | Baseline and Week 4

SECONDARY OUTCOMES:
Sleep Quality: Assessed using the Pittsburgh Sleep Quality Index (PSQI) total score | Baseline and Week 4
General Self-Efficacy: Assessed using the General Self-Efficacy Scale (GSE) score | Baseline and Week 4
Emotional Well-being: Assessed using the World Health Organization Well-being Index (WHO-5) score | Baseline and Week 4
Neck Functional Limitation: Assessed using the Neck Disability Index (NDI) score | Baseline and Week 4
Hand and Shoulder Functionality: Assessed using the Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire score | Baseline and Week 4
Acute Pain Intensity Change: Assessed using the Numerical Rating Scale (NRS) score (0-10) in the specific massage area | Periprocedural
Acute Subjective Well-being Change: Assessed using the Visual Analog Scale (VAS) (0-100 mm) for relaxation, fatigue, and tension | Periprocedural

OTHER OUTCOMES:
Age of Participants | Baseline
  The age of participants calculated from their date of birth. Years
Smoking Status Categories | Baseline
  The classification of participants' smoking status (e.g., Current Smoker, Former Smoker, Never Smoker). Count (Number of Participants per Category)
Body Mass Index (BMI) | Baseline
  Body Mass Index, calculated from weight and height. kg/m2
Duration of Sedentary Work Experience | Baseline
  The total duration of sedentary work experience. Years
Family and Parental Status Categories | Baseline
  The classification of participants based on their family and parental status (e.g., Married, Unmarried, With Children, Without Children). Count (Number of Participants per Category)
Total Physical Activity Level (IPAQ) | Baseline
  Total physical activity level score calculated using the International Physical Activity Questionnaire (IPAQ) short form. Metabolic Equivalent of Task (MET) -minutes/week

IPD SHARING:
Plan to Share IPD: Yes